CLINICAL TRIAL: NCT06684561
Title: EARLY FEASIBILITY STUDY: SAFETY AND EFFICACY OF PHOTON INFUSION SET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Amir Tirosh, Prof. Amir Tirosh, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sheba-24-1530-AT-CTIL
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Infusion sets; insulin pumps; AID system
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): All subjects will be instructed to change the investigational infusion sets (PIS) every 246 hours (10 days & 6 hours) or at set failure. Each subject is required to wear the CGM device continuously.
  defined as any one of the following: After completing 2 sets, the subjects have an optional office visit to download pump and CGM data and will continue to additional two wears. At day 40 or after using 4 completed wears of infusion sets (Note: early infusion set failure with wear time of <6 hours due to insertion failure will be reported, yet not accounted as completed wear), the patients will return to a visit, download pump and CGM data, and end the study.
  if study 1 is successful, participants will enter study 2; , the same study designed will be performed on the current on-market Extended infusion set (EIS) for comparison of clinical performance with the PIS, using the same cohort of pump users
  Interventions: Device: PIS

INTERVENTIONS:
Device: PIS — All subjects will be instructed to change the investigational infusion sets (PIS) every 246 hours (10 days & 6 hours) or at set failure. Each subject is required to wear the CGM device continuously.
  defined as any one of the following: After completing 2 sets, the subjects have an optional office visit to download pump and CGM data and will continue to additional two wears. At day 40 or after using 4 completed wears of infusion sets (Note: early infusion set failure with wear time of <6 hours due to insertion failure will be reported, yet not accounted as completed wear), the patients will return to a visit, download pump and CGM data, and end the study.
  if study 1 is successful, participants will enter study 2; , the same study designed will be performed on the current on-market Extended infusion set (EIS) for comparison of clinical performance with the PIS, using the same cohort of pump users

SUMMARY:
Study 1:

The purpose of this study is to evaluate safety and efficacy of Photon infusion sets (PIS) with new PFAS-free cannula (catheter) in adult patients with Type 1 diabetes for up to 10 days and 6 hours.

This is a 1-center, prospective, open-label, 1-arm study with type 1 patients with diabetes on 780G insulin pump therapy with Guardian™ 4 Continuous Glucose Monitoring (CGM). All subjects will be instructed to change infusion sets every 246 hours (10 days & 6 hours) or at set failure. Each subject is required to wear the CGM device continuously.

After completing 2 sets, the subjects have an optional office visit to download pump and CGM data and will continue to additional two wears. At day 40 or after using 4 completed wears of infusion sets (Note: early infusion set failure with wear time of <6 hours due to insertion failure will be reported, yet not accounted as completed wear), the patients will return to a visit, download pump and CGM data, and end the study.

Photon infusion sets with 6-mm and 9-mm cannula length will be supplied for this study, with selection based on subjects' needs and doctor's recommendation. Subjects will change insulin reservoirs at least every 7 days (the labelled wear duration of the Extended reservoir). The infusion set(s) or reservoir(s) can be replaced independent of each other. The date and time of each infusion set insertion will be recorded in a Daily Log (Diary) which will include the causes of early removal, if occurs.

Study 2: If Study 1 is successful, the same study designed as illustrated in Figure 1 may be performed on the current on-market Extended infusion set (EIS) for comparison of clinical performance with the PIS, using the same cohort of pump users.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes for at least one year
2. Using a MiniMed™ 780G Insulin pump with Guardian sensor
3. Age 18 to 80 years
4. Hemoglobin A1c level less than or equal to 10%
5. Not currently known to be pregnant, nor planning pregnancy during the study.
6. Willingness to follow the protocol and sign the informed consent

Exclusion Criteria:

1. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol.
2. Pregnant or lactating females
3. Subject has Glycosylated hemoglobin (HbA1c)< 10 % at time of screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | 12 months
  The primary outcome is to have no more than 16% of infusion set failures due to "unexplained hyperglycemia" Definition of unexplained hyperglycemia: o The study meter glucose >250 mg/dL (>3 hours post-meal) which may include time during subject's sleeping hours.
  * Failure of a correction dose(s) to lower the study meter glucose by at least 50 mg/dL within 1 hour.
  * One additional correction dose may be given after first correction dose and recommended to use the bolus calculator

IPD SHARING:
Plan to Share IPD: No